CLINICAL TRIAL: NCT05042778
Title: Is Auriculotherapy Responsable for Improvements on Anxiety Students' Prior and After Examinations?
Brief Title: Is Auriculotherapy Responsible for Improvements on Anxiety Students' Prior and After Examinations?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Escola Superior Saúde Santa Maria (Unknown)
Responsible Party: Principal Investigator, Andreia Vieira, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ESSSMUporto
Record Dates: First submitted 2021-08-25; First posted 2021-09-13 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Anxiety
Keywords: Anxiety; Vagus nerve stimulation; auriculotherapy; students
MeSH Terms: conditions — Anxiety Disorders | interventions — Auriculotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auriculotherapy (Experimental): Indwelling fixed semipermanent needles embedded in a skin-colored adhesive tape will be used in active points around the vagus nerve stimulation area.
  Interventions: Other: Auriculotherapy
- No intervention (No Intervention): No auriculotherapy will be applied.

INTERVENTIONS:
Other: Auriculotherapy — A licensed acupuncturist (holder of civil liability insurance) with more than nine years of experience with this technique will apply auriculotherapy. Indwelling fixed semipermanent needles embedded in a skin-coloured adhesive tape will be used at the actives auricular points around the vagus nerve area.
  Arms: Auriculotherapy

SUMMARY:
As the investigators have shown before, there was a tendency for a reduction of anxiety levels on university students after 30 minutes, with auriculotherapy treatment before examinations have started. However, the effect was effective and clinically significant after 48 hours comparing auriculotherapy with placebo and no treatment. In this sense, the investigators intend to perform a new study with a large sample and introduce a new hypothesis. So, this study aims to detect the clinical effect of two auriculotherapy techniques on the anxiety levels of university students.

DETAILED DESCRIPTION:
To treat anxiety, conventional medicine relies on medicines such as benzodiazepines, antidepressants, barbiturates, and antihistamines. However, several authors have reported western medicine cannot resolve all anxiety diseases and the risk of side effects, resistance to pharmacological treatments affects approximately one in three patients with anxiety disorders.

Alternatively, auriculotherapy is a technique similar to reflexology. It is speculated the technique might work in anxiety because groups of pluripotent cells contain information from the whole organism creating regional organization centres representing different parts of the body, through the recruitment of more cortex cells dedicated to specific body areas. Thus reflex points in the ear can incite body responses by the stimulation of reticular formation and the sympathetic and parasympathetic nervous systems. The information that comes from the thermal, Algic and proprioceptive stimuli are transmitted from the auricular pavilion by the fibres of the nerves: trigeminal; Auricular magnum and minor occipital (sensitive branch of the cervical plexus) and the vagus nerve. The vagus nerve is responsible for the parasympathetic innervation of the lung, heart, stomach, and small intestine, as well as the pharynx and larynx muscles and it also sends information to important brain regions (e.g., locus coeruleus, orbitofrontal cortex, hippocampus and at amygdala) in the regulation of anxiety. In turn, the trigeminal nerve controls, mainly, the mastication muscles and the facial sensitivity while the cervical plexus nerve is responsible for neck muscles, diaphragm, and thorax.

ELIGIBILITY:
Inclusion Criteria:

* University students
* Unfamiliar with auriculotherapy,
* No psychological disorders measured through Brief Symptom Inventory scale.

Exclusion Criteria:

* Students having any neurological disease, cardiovascular disease, renal disease or any chronic disease, such as diabetes or hypertension.
* Pregnants.
* Under psychiatric medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Change on Spielberger's State-Trait-Anxiety Inventory (STAI) | Change from baseline to after 8 and 24 hours.
  Was developed by Spielberger and colleagues in 1970, validated for the Portuguese population, with the aim of analyzing anxiety symptoms. STAI is an instrument for measuring the state and trait of anxiety, consisting of two auto-answer questionnaires, each consisting of 20 items. The score ranges from 20 to 80 points on both scales, where 20 to 35 points means not anxious, 36 to 50 points is considered little anxious; 51 to 65 points means moderately anxious; and finally, 66 to 80 points the participant is considered very anxious.
Change on Salivary amylase (U/ml) | Change from baseline to after 16 hours.
  The method responds to both pancreatic and salivary amylase isoenzymes. Samples will be diluted prior to analysis and all measurements are going to be in compliance with the national legal requirements.

SECONDARY OUTCOMES:
Change on Visual analogic scale (VAS) for anxiety | Change from one week before baseline to after 8 and 24 hours.
  Consists of a horizontal or vertical line, 100 mm long, which has marked the classification "totally calm and relaxed" at one end and, at the other, the classification "Worst fear imaginable". The respondent should mark the point that represents the degree of intensity of his anxiety. The distance between the beginning of the line, which corresponds to zero and the marked location, is then measured in centimeters, thus obtaining a numerical classification. The scale is reliable and correlated with STAI-Y1 (p <0.0001) for the level of anxiety and was used on our previous study
Change on quality of sleep | Change from one week before baseline to after 8 and 24 hours.
  The participants will be asked about the quality of sleep during the night before as: 1-no change, 2-better or 3- worse than the quality of sleep during the previous week.
Change on Blood Glucose levels | Change from baseline to after 30 minutes and 24 hours.
  Cortisol acts on two distinct fronts that results in increased amounts of glucose in the bloodstream. It stimulates gluconeogenesis in the liver, and the glucose produced is released into the bloodstream and stored as glycogen. In addition, by potentiating the effects of epinephrine, it elevates glycogenolysis in the liver, thus releasing a large amount of glucose into the bloodstream within minutes.
Test performance | one week after examinations
  After the exam, the test performance (pass or fail) will also be recorded.
Adverse effects | up to one week after baseline
  We will collect data related to auriculotherapy´ adverse effects (e.g, pain, presence of hematoma, vagal reaction, and infection), by replying the Adverse effect questionnaire after the procedure, as well as 1 week after completion of the experimental session.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Machado, Ph.D, Study Director — Instituto de Ciências Biomédicas Abel Salazar
Locations (1):
- ICBAS, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No
Results can be disseminated through workshops or seminars, or newsletters, to reach the largest number of people. Among educational institutions, a workshop can be held on the importance of implementing strategies to reduce situational anxiety. Communications could be whispered at scientific meetings and publications in journals to contribute about auriculotherapy effects, physiologic mechanisms and safety.

REFERENCES:
- [Background] Vieira, A., Hinzmann, M., Silva, K., Santos, M., & Machado, J. (2018). Clinical effect of auricular acupuncture in anxiety levels of students prior to the exams: A randomized controlled trial. European Journal of Integrative Medicine, 20, 188-192. doi:https://doi.org/10.1016/j.eujim.2018.05.012